CLINICAL TRIAL: NCT04425603
Title: Anthology Hip Replacement System - Orthopaedic Data Evolution Panel (ODEP) Surveillance Study
Status: Completed | Type: Observational
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Other Study IDs: R11006-1
Record Dates: First submitted 2020-01-07; First posted 2020-06-11 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Primary Osteoarthritis; Secondary Osteoarthritis; Avascular Necrosis; Primary Total Hip Replacement (THR)
Keywords: THR; Anthology Hip Replacement
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Anthology Hip Replacement System

SUMMARY:
This clinical study will verify the clinical and radiographic performance of the prosthesis when used in human subjects over a period of 10 years. All complications will be documented.

DETAILED DESCRIPTION:
The clinical evaluations will be based on standard, functional and pain parameters Harris Hip Score pre-operatively, and at 6 months, 3, 5, 7.5 and 10 years post-operatively. Postal Oxford questionnaire preoperatively, and yearly thereafter. The objective of this study is to analyse the clinical and radiographic responses and the complication rates for patients undergoing primary total hip arthroplasty using the Anthology Hip Replacement System (Anthology Hip System).

ELIGIBILITY:
Inclusion criteria:

1. Those presenting with primary or secondary osteoarthritis or avascular necrosis of the femoral head or patients suitable for a primary total hip replacement. This is the patient group that will benefit from operative surgery to treat osteoarthritis.
2. Those deemed capable of giving informed consent, understanding the aims of the study and expressing willingness to comply with the post-operative review programme. Patients capable of giving informed consent are eligible for inclusion into the study.
3. Participants who signed the Ethics Committee approved specific Informed Consent Form prior to surgery. Patients who have not given informed consent will not be eligible for inclusion into the study.

Exclusion criteria:

1. Patients whose prospects for a recovery to independent mobility would be compromised by known coexistent, medical problems.
2. Patients not suitable for primary hip replacement.
3. Patients with active or suspected infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Those presenting with primary or secondary osteoarthritis or avascular necrosis of the femoral head or patients suitable for a primary total hip replacement (THR).
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2007-04-30 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score - 10 years | 10 years post operative
  The Harris Hip Score is a joint specific score that consists of 10 items covering domains of pain (1 item, 0-44 points), function (7 items, 0-47 points), functional activities, absence of deformity (1 item, 0 or 4 points), and hip range of motion (2 items, 0-5 points). Scores range from 0 (worst) to 100 (best).
Quality of life with Oxford Hip Score (postal) - 10 years | 10 years post operative
  Patients are asked to reflect on their pain and functional ability over the previous four weeks. There are two domains (pain and function) with six items or questions in each. Each item has five possible responses. In the original scoring responses were from 1 = least difficult to 5= most difficult. Item scores are summed to give a total score from anywhere between 12 and 60. The lower the score, the better the outcome.
Quality of life with EuroQol Questionnaire (EQ-5D) -10 years | 10 years post operative
  The descriptive system consists of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which takes one of three responses. The responses record three levels of severity (no problems/some or moderate problems/extreme problems) within a particular dimension. The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. This information can be used as a quantitative measure of health outcome as judged by the individual respondents.

SECONDARY OUTCOMES:
Harris Hip Score | Pre-operative and 6 months, 3 years, 5 years, and 7.5 years post operative
  The Harris Hip Score is a joint specific score that consists of 10 items covering domains of pain (1 item, 0-44 points), function (7 items, 0-47 points), functional activities, absence of deformity (1 item, 0 or 4 points), and hip range of motion (2 items, 0-5 points). Scores range from 0 (worst) to 100 (best).
Quality of life with Oxford Hip Score (postal) | Pre-operative and 6 months, 3 years, 5 years, and 7.5 years post operative
  Patients are asked to reflect on their pain and functional ability over the previous four weeks. There are two domains (pain and function) with six items or questions in each. Each item has five possible responses. In the original scoring responses were from 1 = least difficult to 5= most difficult. Item scores are summed to give a total score from anywhere between 12 and 60. The lower the score, the better the outcome.
Quality of life with EuroQol Questionnaire (EQ-5D) | Pre-operative and 6 months, 3 years, 5 years, and 7.5 years post operative
  The descriptive system consists of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which takes one of three responses. The responses record three levels of severity (no problems/some or moderate problems/extreme problems) within a particular dimension. The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. This information can be used as a quantitative measure of health outcome as judged by the individual respondents.
Device-related complications | 6 months, 3 years, 5 years, 7.5 years, and 10 years post operative
  Complications and adverse events will be noted at each follow-up and using clinical judgement it will be determined whether the event is device related
Number of revisions or withdrawals for any reason | 6 months, 3 years, 5 years, 7.5 years, and 10 years post operative
Radiographic evaluations | Pre-operative, peri-operative, 6 months, 3 years, 5 years, 7.5 years, and 10 years post operative
  Anterior-posterior, and lateral view x-rays of the femur and pelvis of the affected hip will be evaluated. X-rays will be reviewed and specific information regarding presence/absence/location of radiolucent lines and implant positions and alignment will be recorded.
Survival Rate | 10 years post operative
  The survival rate will be calculated according to the method in accordance with Kaplan-Meier stating the 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Field, MD, Principal Investigator — South West London Elective Orthopaedic Centre (SWLEOC); Helmut Zahn, MD, Principal Investigator — William Harvey Hospital East Kent NHS Trust; Pankaj Sharma, MD, Principal Investigator — Ashford and St. Peter's NHS Trust; Tony Andrade, MD, Principal Investigator — Royal Berkshire NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - William Harvey Hospital East Kent NHS Trust, Ashford
  - Ashford and St. Peter's NHS Trust, Chertsey
  - South West London Elective Orthopaedic Centre (SWLEOC), Epsom
  - Royal Berkshire NHS Foundation Trust, Reading

IPD SHARING:
Plan to Share IPD: No